CLINICAL TRIAL: NCT02391103
Title: Effects of Neuromuscular Electrical Stimulation on Muscle Mass and Strength in Critically Ill Patients After Cardiothoracic Surgery. An Ultrasound-Based Randomized Controlled Trial
Brief Title: Effects of Neuromuscular Electrical Stimulation on Muscle Mass and Strength in Critically Ill Patients After Cardiothoracic Surgery
Acronym: Catastim 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Arabella Fischer, MD, resident, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1072/2010
Record Dates: First submitted 2015-03-07; First posted 2015-03-18 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Neuromuscular Electrical Stimulation; Intensive Care Unit Acquired Weakness; Muscle Wasting; Muscle Loss
MeSH Terms: conditions — Muscular Atrophy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- NMES group (Experimental): Anterior muscles of both thighs were electrically stimulated twice a day (2×30 minutes of NMES with a break of at least 30 minutes between both sessions) 7 days a week during the entire ICU stay but no longer than 14 days, starting on postoperative day 1. Highest tolerable intensity was applied.
  Interventions: Device: Compex 3 Professional (CefarCompex Medical AB) stimulator
- Control group (Sham Comparator): In the control group, the electrodes were applied, connected to the stimulator, but no electricity was delivered.
  Interventions: Device: sham-stimulation

INTERVENTIONS:
Device: Compex 3 Professional (CefarCompex Medical AB) stimulator — NMES
  Arms: NMES group
Device: sham-stimulation — no electricity applied
  Arms: Control group

SUMMARY:
The purposes of this study are 1) to determine whether neuromuscular electrical stimulation (NMES) is effective in preventing loss of muscle mass and strength and 2) to observe the time variation of MLT and strength from preoperative day to hospital discharge.

DETAILED DESCRIPTION:
In the amendment of June 2011, a twofold study setting was defined in order to recruit patients not only before, but also after cardiothoracic surgery. In sample A, patients were recruited before surgery. In sample B, patients were recruited after surgery. On postoperative day 1, randomization was performed for sample A and B separately. To ensure balance of the NMES and control groups with respect to disease severity, randomization was stratified by the SAPS II score on the first postoperative day. In the intervention group, the anterior muscles of both thighs were electrically stimulated from the first postoperative day until ICU discharge for a maximum of 14 days. In the control group, the electrodes were applied, but no electricity was delivered.The primary outcomes muscle layer thickness (MLT) and muscle strength were assessed from the first postoperative day to ICU discharge and at hospital discharge. All patients in sample A had an additional assessment of MLT and strength before surgery.

All data are analyzed according to the intention-to-treat principle with no imputation for any missing data. Linear mixed models are used to account for the repeated measurements per patient and to determine any fixed effects on MLT and MRC score.

ELIGIBILITY:
Inclusion Criteria:

* patients before/after cardiothoracic surgery
* ICU stay > 48 hours

Exclusion Criteria:

* body mass index > 40 kg/m2
* severe leg swelling
* implanted ventricular assist device (RVAD, LVAD, BiVAD)
* implanted intra-aortic balloon pump (IABP)
* neuromuscular diseases
* skin lesions in stimulation area
* leg excluded if implant (hip or knee replacement) in stimulation area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2011-05; Primary Completion 2012-07 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Muscle layer thickness (MLT) | on preoperative day, from postoperative day 1 onwards every other ICU day for the duration of the ICU stay (expected average of ICU stay: 7 days) and at day of hospital discharge (expected average of hospital stay: 20 days)
  Muscle layer thickness of the anterior muscles of the thigh using two-dimensional B-mode ultrasound
Muscle strength | on preoperative day, from postoperative day 1 onwards every day for the duration of the ICU stay (expected average of ICU stay: 7 days), at day of hospital discharge (expected average of hospital stay: 20 days)
  Muscle strength using Medical Research Council (MRC) score and hand dynamometry

SECONDARY OUTCOMES:
JAGS score | on preoperative day, on day of ICU discharge (expected average of ICU stay: 7 days), on day of hospital discharge (expected average of hospital stay: 20 days)
  JAGS score
Timed Up and Go test | on preoperative day, on day of hospital discharge (expected average of hospital stay: 20 days)
  Timed Get Up and Go test
FIM score | on preoperative day, on day of hospital discharge (expected average of hospital stay: 20 days)
  Functional Independance Measure (FIM) score
SF-12 score | on preoperative day, on day of hospital discharge (expected average of hospital stay: 20 days)
  12-item Short Form Health Survey (SF-12)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hiesmayr, MD, Prof., Study Director — Medical University of Vienna; Arabella Fischer, MD, Principal Investigator — Medical University of Vienna

REFERENCES:
- [Background] Gerovasili V, Stefanidis K, Vitzilaios K, Karatzanos E, Politis P, Koroneos A, Chatzimichail A, Routsi C, Roussos C, Nanas S. Electrical muscle stimulation preserves the muscle mass of critically ill patients: a randomized study. Crit Care. 2009;13(5):R161. doi: 10.1186/cc8123. Epub 2009 Oct 8. PMID 19814793
- [Background] Hirose T, Shiozaki T, Shimizu K, Mouri T, Noguchi K, Ohnishi M, Shimazu T. The effect of electrical muscle stimulation on the prevention of disuse muscle atrophy in patients with consciousness disturbance in the intensive care unit. J Crit Care. 2013 Aug;28(4):536.e1-7. doi: 10.1016/j.jcrc.2013.02.010. Epub 2013 Apr 3. PMID 23561945
- [Background] Rodriguez PO, Setten M, Maskin LP, Bonelli I, Vidomlansky SR, Attie S, Frosiani SL, Kozima S, Valentini R. Muscle weakness in septic patients requiring mechanical ventilation: protective effect of transcutaneous neuromuscular electrical stimulation. J Crit Care. 2012 Jun;27(3):319.e1-8. doi: 10.1016/j.jcrc.2011.04.010. Epub 2011 Jun 28. PMID 21715139
- [Background] Kho ME, Truong AD, Zanni JM, Ciesla ND, Brower RG, Palmer JB, Needham DM. Neuromuscular electrical stimulation in mechanically ventilated patients: a randomized, sham-controlled pilot trial with blinded outcome assessment. J Crit Care. 2015 Feb;30(1):32-9. doi: 10.1016/j.jcrc.2014.09.014. Epub 2014 Sep 22. PMID 25307979
- [Background] Abdellaoui A, Prefaut C, Gouzi F, Couillard A, Coisy-Quivy M, Hugon G, Molinari N, Lafontaine T, Jonquet O, Laoudj-Chenivesse D, Hayot M. Skeletal muscle effects of electrostimulation after COPD exacerbation: a pilot study. Eur Respir J. 2011 Oct;38(4):781-8. doi: 10.1183/09031936.00167110. Epub 2011 Feb 24. PMID 21349913
- [Background] Routsi C, Gerovasili V, Vasileiadis I, Karatzanos E, Pitsolis T, Tripodaki E, Markaki V, Zervakis D, Nanas S. Electrical muscle stimulation prevents critical illness polyneuromyopathy: a randomized parallel intervention trial. Crit Care. 2010;14(2):R74. doi: 10.1186/cc8987. Epub 2010 Apr 28. PMID 20426834
- [Background] Zanotti E, Felicetti G, Maini M, Fracchia C. Peripheral muscle strength training in bed-bound patients with COPD receiving mechanical ventilation: effect of electrical stimulation. Chest. 2003 Jul;124(1):292-6. doi: 10.1378/chest.124.1.292. PMID 12853536
- [Background] Puthucheary ZA, Phadke R, Rawal J, McPhail MJ, Sidhu PS, Rowlerson A, Moxham J, Harridge S, Hart N, Montgomery HE. Qualitative Ultrasound in Acute Critical Illness Muscle Wasting. Crit Care Med. 2015 Aug;43(8):1603-11. doi: 10.1097/CCM.0000000000001016. PMID 25882765
- [Background] Puthucheary ZA, Rawal J, McPhail M, Connolly B, Ratnayake G, Chan P, Hopkinson NS, Phadke R, Dew T, Sidhu PS, Velloso C, Seymour J, Agley CC, Selby A, Limb M, Edwards LM, Smith K, Rowlerson A, Rennie MJ, Moxham J, Harridge SD, Hart N, Montgomery HE. Acute skeletal muscle wasting in critical illness. JAMA. 2013 Oct 16;310(15):1591-600. doi: 10.1001/jama.2013.278481. PMID 24108501
- [Derived] Fischer A, Spiegl M, Altmann K, Winkler A, Salamon A, Themessl-Huber M, Mouhieddine M, Strasser EM, Schiferer A, Paternostro-Sluga T, Hiesmayr M. Muscle mass, strength and functional outcomes in critically ill patients after cardiothoracic surgery: does neuromuscular electrical stimulation help? The Catastim 2 randomized controlled trial. Crit Care. 2016 Jan 29;20:30. doi: 10.1186/s13054-016-1199-3. PMID 26825278